CLINICAL TRIAL: NCT05463627
Title: Effects of Metformin on Metabolic and Reproductive Outcomes in Chinese PCOS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2021-184-B
Record Dates: First submitted 2022-03-24; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-03

CONDITIONS: Polycystic Ovary Syndrome; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BMI<24 kg/m2: women diagnosed with PCOS with BMI<24 kg/m2
  Interventions: Drug: Metformin
- BMI24-28 kg/m2: women diagnosed with PCOS with BMI24-28 kg/m2
  Interventions: Drug: Metformin
- BMI>28 kg/m2: women diagnosed with PCOS with BMI>28kg/m2
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — All participants among the three groups were treated with metformin
  Other Names: melbine

SUMMARY:
Polycystic ovary syndrome (PCOS) is a reproductive endocrine disease characterized by reproductive and metabolic abnormalities, which is a crucial cause of female infertility and an essential risk factor for type 2 diabetes. At present, there exist several clinical trials and studies on the usage of metformin in the treatment of PCOS patients in prediabetes, and the practical application of metformin in clinical practice has years of history. The treatment plan of metformin is of great significance in preventing type 2 diabetes in PCOS patients and assisting pregnancy in PCOS infertile patients.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a real world study on effects of metformin on the improvement of metabolism and reproductive outcome in Chinese prediabetic PCOS patients by collecting relevant medical system records from Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine as real world data and a significant supplement to clinical trial studies. At the same time, obese and non-obese PCOS patients may have different mechanisms of insulin resistance, so this study stratified PCOS patients to analyze whether metformin can improve treatment results for PCOS patients with prediabetes according to different body mass index (BMI).The investigator's study is the first real world study to investigate Chinese pre-diabetes PCOS patients treated by metformin and the metabolic and reproductive outcomes, which is innovative. The investigator's research also has a guiding significance for the practical application of metformin in improving glucose metabolism and reproductive outcomes in patients with different body weight in clinical practice, and has great relevance for PCOS patients to reduce long-term complications and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Females at the age of 18-45years old;
2. Diagnosed with PCOS or/and impaired glucose regulation (IGR)/diabetes(DM)
3. Metformin regimens were used without other metabolic agents
4. The diagnosis of PCOS is based on the 2003 Rotterdam criteria and the diagnostic criteria for impaired glucose regulation (IGR) and type 2 diabetes are based on the 2021 American Diabetes Association(ADA) diagnosis criteria.

Exclusion Criteria:

1. Severe liver and kidney dysfunction (ALT is greater than 2.5 times the upper limit of normal, or Cr>132umol/l, or eGFR <60 mL/min/1.73m2), psychosis, accompanied by severe infection, severe anemia, neutropenia disease;
2. Participated in clinical trials of other drugs within 3 months;
3. In the past 5 years, there have been treated or untreated organ system tumors (except local skin basal cell carcinoma), regardless of whether there is evidence of local recurrence or metastasis;
4. A history of psychoactive substance abuse, including alcohol and a history of alcohol-related illnesses in the past 2 years;
5. Any conditions judged by the investigator that affect enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese,overweight and normal-weight women aged 18-45 years (in childbearing age)with PCOS or/and IGR/DM were expected enrolled in our study
Sampling Method: Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Reversed insulin resistance or restored glucose homeostasis in women with PCOS | 5 years
  Compared with the baseline in three groups, the rate of reversed insulin resistance or restored glucose homeostasis

SECONDARY OUTCOMES:
change in the level of BMI | 5 years
  Compared with the baseline in three groups, the level of BMI is one of the metabolic index to evaluate metabolic outcome
change in the level of glycated hemoglobin(HbA1c) | 5 years
  Compared with the baseline in three groups, the level of HbA1c is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of 0'-180'Plasma Glucose(PG) | 5 years
  Compared with the baseline in three groups, the level of 0'-180'PG from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of 0'-180'insulin(ins) | 5 years
  Compared with the baseline in three groups, the level of 0'-180'ins from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of 0'-180'C-Peptide | 5 years
  Compared with the baseline in three groups, the level of 0'-180'C-Peptide from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of β cell homeostatic model assessment(HOMA-β) | 5 years
  Compared with the baseline in three groups, the level of HOMA-β calculated from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of Matsuda Index(MI) | 5 years
  Compared with the baseline in three groups, the level of MI calculated from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of deposition index(DI) | 5 years
  Compared with the baseline in three groups, the level of DI calculated from oral glucose tolerance test is one of the metabolic index to evaluate glucose metabolic outcome
change in the level of waist-hip ratio(WHR) | 5 years
  Compared with the baseline in three groups, the level of WHR is one of the metabolic index to evaluate metabolic outcome
change in the level of Luteinizing hormone(LH) | 5 years
  Compared with the baseline in three groups, the level of LH is one of the metabolic index to evaluate Reproductive outcome
change in the level of Follicle stimulating hormone(FSH) | 5 years
  Compared with the baseline in three groups, the level of FSH is one of the metabolic index to evaluate Reproductive outcome
change in the level of Prolactin(PRL) | 5 years
  Compared with the baseline in three groups, the level of PRL is one of the metabolic index to evaluate Reproductive outcome
change in the level of estradiol(E2) | 5 years
  Compared with the baseline in three groups, the level of E2 is one of the metabolic index to evaluate Reproductive outcome
change in the level of testosterone(T) | 5 years
  Compared with the baseline in three groups, the level of T is one of the metabolic index to evaluate Reproductive outcome
change in the level of Sex hormone-binding globulin(SHBG) | 5 years
  Compared with the baseline in three groups, the level of SHBG is one of the metabolic index to evaluate Reproductive outcome
change in the level of Dehydroepiandrosterone sulfate(DHEAS) | 5 years
  Compared with the baseline in three groups, the level of DHEAS is one of the metabolic index to evaluate Reproductive outcome
change in the level of Androstenedione(A2) | 5 years
  Compared with the baseline in three groups, the level of A2 is one of the metabolic index to evaluate Reproductive outcome
pregnancy rate | 5 years
  Compared with the baseline in three groups, pregnancy rate is one of the index to evaluate Reproductive outcome
live birth rate | 5 years
  Compared with the baseline in three groups, live birth rate is one of the index to evaluate Reproductive outcome
improvement rate of menstrual cycle | 5 years
  Compared with the baseline in three groups, improvement rate of menstrual cycle is one of the index to evaluate Reproductive outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, Dr., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen AJT, Stage TB, Glintborg D, Andersen M, Christensen MMH. The Pharmacogenetics of Metformin in Women with Polycystic Ovary Syndrome: A Randomized Trial. Basic Clin Pharmacol Toxicol. 2018 Feb;122(2):239-244. doi: 10.1111/bcpt.12874. Epub 2017 Sep 19. PMID 28834135
- [Background] Li Y, Tan J, Wang Q, Duan C, Hu Y, Huang W. Comparing the individual effects of metformin and rosiglitazone and their combination in obese women with polycystic ovary syndrome: a randomized controlled trial. Fertil Steril. 2020 Jan;113(1):197-204. doi: 10.1016/j.fertnstert.2019.09.011. Epub 2019 Nov 9. PMID 31718828
- [Background] Xiong F, Xiao J, Bai Y, Zhang Y, Li Q, Lishuang X. Metformin inhibits estradiol and progesterone-induced decidualization of endometrial stromal cells by regulating expression of progesterone receptor, cytokines and matrix metalloproteinases. Biomed Pharmacother. 2019 Jan;109:1578-1585. doi: 10.1016/j.biopha.2018.10.128. Epub 2018 Nov 15. PMID 30551411